CLINICAL TRIAL: NCT06681961
Title: The Therapeutic Effects of a Dynamics Closed Kinetic Chain Exercise Combination With Hip Adduction in Patients With Patellofemoral Pain Syndrome
Brief Title: Effects of a Squatting With Hip Adduction in Patients With Patellofemoral Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Wei-Hsien Hong, China Medical University, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMUH106-REC1-014
Record Dates: First submitted 2024-11-04; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: PFPS
Keywords: Patellofemoral pain syndrome; Vastus medialis obliquus; Squatting; Hip adduction
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Population Groups

STUDY DESIGN:
Intervention Model Description: Thirty PFPS participants were randomly assigned to conventional squatting (SQU) (n=15) or squatting with hip adduction (SQU-HA) (n=15) groups. Participants were blinded to the interventions used in the other group.
Who Masked: Participant
Masking Description: This was a prospective, randomized-controlled trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- squatting with hip adduction (SQU-HA) group (Experimental): The participants stood equally on both legs on the floor with their feet shoulder-width apart and angled outward at 20°-30°. After a warm-up, the participants performed 45° squats with squeezing a Swiss ball of 18-cm diameter at a slow speed of 2 s for flexion and extension from the standing posture by using a commercial metronome. The squatting with knee flexion from 0° to 45° was the safest for people with PFPS.
  Interventions: Other: squatting with hip adduction (SQU-HA) group
- squatting (SQU) group (Other): The participants stood equally on both legs on the floor with their feet shoulder-width apart and angled outward at 20°-30°. After a warm-up, the participants performed 45° squats at a slow speed of 2 s for flexion and extension from the standing posture by using a commercial metronome. The squatting with knee flexion from 0° to 45° was the safest for people with PFPS.
  Interventions: Other: squatting with hip adduction (SQU-HA) group

INTERVENTIONS:
Other: squatting with hip adduction (SQU-HA) group — The intervention comprised three sets of 15 repetitions with resting 5-min between sets, followed by IT band stretching for five repetitions. Each participant performed the respective exercise 5 days a week, with 2 days of rest, for 8 weeks.
  Other Names: squatting (SQU) group

SUMMARY:
An imbalance in the activation and onset time of the vastus medialis oblique (VMO) and vastus lateralis (VL) muscles may be one of the primary causes of PFPS. Several studies have discussed various exercise methods believed to selectively contract the (VMO) muscle for treating patellofemoral pain syndrome. VMO activity is higher during static closed-chain tasks combined with hip adduction, indicating that performing hip adduction exercises may selectively strengthen the VMO muscle.

DETAILED DESCRIPTION:
Patellofemoral pain syndrome (PFPS) poses challenges in motor control and pain management, especially regarding balanced muscle activation of the vastus medialis oblique (VMO) and vastus lateralis (VL). This study introduces a home-based PFPS rehabilitation approach involving a squat exercise program with hip adduction, examining its effects on motor control and clinical outcomes. Thirty PFPS participants were randomly assigned to conventional squatting (SQU) or squatting with hip adduction (SQU-HA) groups. Participants performed exercises five days a week for 8 weeks, with pre- and post-assessments capturing clinical measures and motor control indicators using electromyography (EMG). This home-based program, integrating hip adduction into squats, enhances motor control, reduces knee stress, and improves daily function, ensuring continued care post-pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-50 years.
* Pain around the patella at least two of the following activities¬-standing up after prolonged sitting, going up and down the stairs, running, jumping, squatting, kneeling, and high-angle knee flexion for a long time.
* Knee joint pain for ≥3 months.
* Pain level of ≥ 30 mm on a 100-mm visual analog scale (VAS).

Exclusion Criteria:

* Had a history of patellar subluxation, dislocation, or knee surgery.
* Had central or peripheral neurological pathology.
* Had an obvious knee joint deformity or lower extremity malalignment.
* Experienced severe knee joint pain (VAS) score > 80 mm), or received nonsteroidal anti-inflammatory drugs, injections, or physical therapy within the past 3 months.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-01-05 (Actual)

PRIMARY OUTCOMES:
Amplitudes of muscle activation (unit: %MVC) | pre-intervention and after 8-week intervention
  represented the mean RMSs for each muscle which was normalized by the maximal voluntary contractions (MVC).
VMO/VL ratio | pre-intervention and after 8-week intervention
  represents the amplitude ratio of VMO relative to VL.
Onset time (unit: msec) | pre-intervention and after 8-week intervention
  at 200 ms before the beginning of the trial, as the baseline, the onset of EMG activation was identified as the point at which the EMG amplitude was more than three standard deviations from the baseline level for at least 25 ms.
VMO - VL (unit: msec) | pre-intervention and after 8-week intervention
  represented the onset time differences of VMO relative to VL, with a positive (negative) value indicating a delayed (early) onset time of VMO relative to VL.
Q angle (unit: degree) | pre-intervention and after 8-week intervention
  The angle was calculated with the intersection formed by two lines crossing the center of the patella. The first line went from the ASIS to the center of the patella and the second from the anterior tuberosity of the tibia to the center of the patella.
The visual analogue scale (VAS) (unit: mm) | pre-intervention and after 8-week intervention
  VAS was used to assess pain severity. The participants were asked to mark their pain levels on a 100-mm ruler (ranging from 0 = "no pain" to 100 = "unbearable pain") before and after the exercise program.
patellofemoral pain severity scale (PSS) (unit: score) | pre-intervention and after 8-week intervention
  PSS was used to measure PFPS associated with functional activities over the past week. The scale comprises 10 items, including climbing/descending stairs, squatting, walking, jogging, running/sprinting, participating in a sport, sitting with knees bent (for 20 min), kneeling, resting, and following an activity. The maximum score was 100 points. The participants rated their pain on a 100-mm VAS, ranging from 0 = "no pain" to 100 = "unbearable pain".

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Hsien Hong, PhD, Principal Investigator — China Medical University, Taiwan
Locations (1):
- China Medical University, Taichung, Taiwan